CLINICAL TRIAL: NCT04496362
Title: Single Center Open Label Randomized Study Evaluating Safety and Efficacy of Subcutaneous Heparin Compared to Standard of Care Intravenous Heparin Anticoagulation During Veno-venous Extracorporeal Membrane Oxygenation for Respiratory Failure
Brief Title: Veno-venous Extracorporeal Membrane Oxygenation (VV-ECMO) Heparin Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 018-543
Record Dates: First submitted 2020-07-13; First posted 2020-08-03 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: ECMO; Heparin; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- subcutaneous heparin anticoagulation (Experimental): Experimental arm
  Interventions: Drug: subcutaneous heparin anticoagulation
- systemic intravenous anticoagulation (No Intervention): SOC arm

INTERVENTIONS:
Drug: subcutaneous heparin anticoagulation — The primary objective of this study is to evaluate the safety and efficacy of subcutaneous heparin anticoagulation compared to the standard of care systemic intravenous anticoagulation during veno-venous extracorporeal membrane oxygenation for respiratory failure. Subjects will be prospectively randomized in 1:1 ratio to subcutaneous heparin anticoagulation or systemic intravenous anticoagulation and followed until 1 week after discontinuation from ECMO support.
  Other Names: systemic intravenous anticoagulation as SOC
  Arms: subcutaneous heparin anticoagulation

SUMMARY:
This single-center, open-label study will evaluate the safety and efficacy of subcutaneous heparin anticoagulation compared to the standard of care systemic intravenous anticoagulation during veno-venous extracorporeal membrane oxygenation for respiratory failure.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) has been increasing used over the past decade as supportive therapy in patients with respiratory failure, in order to avoid life-threatening hypoxemia, in cases otherwise refractory to conventional treatment. Veno-venous ECMO (VV ECMO) removes carbon dioxide and significantly improves oxygenation in patients with severe lung failure. System anticoagulation is provided for patients undergoing ECMO therapy to prevent clot formation in the ECMO circuit cannulas, circuit tubing, centrifugal pump, and/or oxygenator. Heparin is the standard anticoagulant for ECMO therapy.

Although technological advancements and increasing clinical experience have made the use of VV ECMO safer, bleeding and thrombosis are common complications accounting for the majority of morbidity and mortality in ECMO-treated patients.The optimal anticoagulation management for patients on VV ECMO is not known. Thrombotic episodes, characterized mainly by circuit-related clotting, have become more manageable with improvements in ECMO circuit technology and heparin-coated lines.

The Extracorporeal Life Support Organization (ELSO) guidelines describe bleeding as the most common complication during extracorporeal life support. Bleeding has been reported to occur in as many as 30% of patients receiving ECMO therapy, and depending on the site of the hemorrhagic complication, can be fatal. Bleeding may occur from mucous membranes, the uterus in women in childbearing years, the GI tract, or bleeding into the head or brain parenchyma. Intra-cranial hemorrhage is the most serious and usually extensive and fatal complication.Intra-cranial hemorrhage was identified in more than 40% of non-survivors treated with ECMO during the H1N1 flu outbreak of 2009. Other less serious complications associated with anticoagulation are anemia and the risks associated with transfusions. Review of our own institutional ECMO experience revealed 10 cases of VV ECMO during which anticoagulation had to be held for clinical reasons, all without subsequent increases in thrombotic complications.

Identifying the safest approach to anticoagulation is essential to the future management of patients on ECMO support. In this prospective randomized clinical trial, the investigators propose to evaluate the safety and efficacy of subcutaneous heparin anticoagulation compared to the standard of care systemic intravenous anticoagulation in subjects requiring veno-venous extracorporeal membrane oxygenation for respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Respiratory failure requiring VV-ECMO support
3. Subject or appointed health care proxy/LAR is able to understand and sign the informed consent form

Exclusion Criteria:

1. Subject currently enrolled in another interventional research trial
2. History of hypersensitivity/adverse reaction to heparin
3. Proven Heparin induced thrombocytopenia (HIT)
4. History of patent foramen ovale (PFO)
5. Recent surgery or other contraindication to systemic anticoagulation, e.g. intracranial bleed
6. Medical indication other than ECMO for systemic anticoagulation, e.g. pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of bleeding complication | 1 week
  Safety will be assessed by incidence of bleeding complication (clinically apparent or need for blood transfusion without identified source)
Incidence of thrombotic complications requiring intervention | 1 week
  Safety will be assessed by incidence of thrombotic complications requiring intervention (initiation of systemic anticoagulation or oxygenator exchange)
Incidence of deep venous thrombosis | 1 week
  Incidence of deep venous thrombosis as assessed by four extremity venous ultrasound at one week post-decannulation

SECONDARY OUTCOMES:
Mortality | 1 year
  Directly related to bleeding and clotting

CONTACTS AND LOCATIONS:
Overall Officials: Gary Schwartz, MD, Principal Investigator — BSWH
Locations (1):
- Baylor Scott & White Health research institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data (IPD)

REFERENCES:
- [Background] Sklar MC, Sy E, Lequier L, Fan E, Kanji HD. Anticoagulation Practices during Venovenous Extracorporeal Membrane Oxygenation for Respiratory Failure. A Systematic Review. Ann Am Thorac Soc. 2016 Dec;13(12):2242-2250. doi: 10.1513/AnnalsATS.201605-364SR. PMID 27690525
- [Background] Vaugh N, Hernandez O, Estroff J. Extracorporeal Membrane Oxygenation without Anticoagulation in Traumatic Brain Injury. Poster Presentation, American College of Surgeons Texas Chapter State Meeting, February 23-25, 2017, Austin, TX.
- [Background] Aubron C, DePuydt J, Belon F, Bailey M, Schmidt M, Sheldrake J, Murphy D, Scheinkestel C, Cooper DJ, Capellier G, Pellegrino V, Pilcher D, McQuilten Z. Predictive factors of bleeding events in adults undergoing extracorporeal membrane oxygenation. Ann Intensive Care. 2016 Dec;6(1):97. doi: 10.1186/s13613-016-0196-7. Epub 2016 Oct 6. PMID 27714705
- [Background] ELSO Guidelines for Adult Respiratory Failure August, 2017.